CLINICAL TRIAL: NCT04747223
Title: Step Rate Retraining to Reduce Injury and Disability: A Randomized Controlled Trial
Brief Title: Step Rate Retraining to Reduce Injury and Disability (STRIDe)
Acronym: STRIDe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Army-Baylor University Doctoral Program in Physical Therapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C.2020.058d
Record Dates: First submitted 2020-07-24; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Overuse Injury; Lower Extremity Problem; Stress Injury, Repetitive; Patellofemoral Pain Syndrome; Shin Splint
Keywords: Running-related lower extremity overuse injuries
MeSH Terms: conditions — Cumulative Trauma Disorders; Patellofemoral Pain Syndrome; Medial Tibial Stress Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants are masked to group assignment. Investigators are blinded to participant's group at follow-ups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retraining (RT) Group (Experimental): The retraining group will receive a watch accelerometer to use for monitoring their step rate with instructions to increase their preferred step rate by 7.5% over the ten in-field training sessions.
  Interventions: Other: Run Gait Retraining
- Control (CON) Group (No Intervention): The control group will receive the same device to monitor their pace but receive no instruction to change their preferred step rate over the ten in-field training sessions.

INTERVENTIONS:
Other: Run Gait Retraining — Running step rate will be retrained by real-time biofeedback via a watch accelerometer. Recent literature showed that performing gait retraining by altering step rate reduces loading rates and joint stress that are associated with lower extremity injuries (Wilson et al 2014, Lenhart et al 2014, Heidersheit et al 2011).
  Arms: Retraining (RT) Group

SUMMARY:
This study will be the first project to evaluate the effectiveness of wearable technology (Garmin Forerunner35) while performing gait retraining in field on military members. The watch will provide real time feedback to the runner on their step rate while performing running sessions outside of the lab. This allows the runner to modify their step rate to meet a recommended step rate provided by the study team member.

Aim 1: To demonstrate the utility of wearable sensors to modify running step rate through real time biofeedback.

Aim 2: To determine whether altering step rate using real time biofeedback reduces lower extremity musculoskeletal injury reoccurrence within 1 year post training.

DETAILED DESCRIPTION:
Volunteers meeting all inclusion and exclusion criteria will read and sign an informed consent form approved by the institutional review board (IRB). After consenting, each participant will answer a demographic questionnaire related to injury history and pertinent injury risk factors (location, duration and type of previous injury, profile time, height, weight, changes in menstruation, etc). The participant will then undergo a running analysis in which the individual will run on an instrumented treadmill while video of running form in the sagittal plane and frontal plane are captured using two stationary two-dimensional digital cameras sampling at 240 Hz. The video will capture the runner from the waist down in order to protect privacy and blinding. Information collected from the treadmill will include AVLR of vGRF, while step rate and other kinematic information will be collected from video analysis. Volunteers will run at their self-selected pace for three minutes on a treadmill, with step rate and AVLR analyzed during the last minute of running. During the inital data collection, if the participant's step rate is greater than 176 spm, the participant will be exluded from the study at this time. The same data collection procedure will be repeated for all participants after retraining and for a subset of participants at 6 months to observe post intervention AVLR and step rate.

Volunteers will then be placed into a retraining group and a control group through random allocation. Each participant, regardless of group, will be provided a Garmin Forerunner35 to use while performing PRT with their unit and/or personal physical training for ten in-field training sessions. The ten in-field training sessions will be performed by the participant outside of the researcher's lab without a researcher present. The participant will be instructed to return to their normal running routine, but to use the watch during 10 running sessions to either monitor and modify their step rate for the retraining group or their pace and distance for the control group. Both groups will receive a training log to track their training sessions.

The retraining group will receive a watch accelerometer to use for monitoring their step rate with instructions to increase their preferred step rate by 7.5% over the ten in-field training sessions. The runner will receive a training log with a target step rate recorded on it. The target step rate will be a 7.5% increase from the preferred step rate the runner used during the gait analysis. The researcher will provide instruction to the participant to match the target step rate while the participants are performing their in-field training sessions by using the watch to monitor their step rate. The watch provides the runner with real-time feedback on their step rate. This allows the runner to monitor their step rate while running and the runner should either increase or decrease their step rate to meet the target step rate provided by the study team member. Training units at FT. Sam Houston perform ability group or self-paced runs for the majority of their endurance training, so participants should not have difficulty adjusting their step rates IAW study plans. Willy et al. was successful using eight in-field training sessions to sustain a 7.5% increase in step rate 1 month post-training in healthy runners (Willy 2016). Adherence to step rate will be assessed at the follow-up by reviewing the last 7 training sessions in the history of the watch. The watch only saves 7 sessions at a time to the watch memory without connecting to an internet database. Viewing the last 7 sessions allows the investigators to assess adherence without relying on the runner to upload data to a server before the participants have completed their training sessions. The average step rate from the last 7 training sessions will be input into an excel spreadsheet and the training sessions will be deleted from the watch.

The control group will receive the same device to monitor their pace but receive no instruction to change their preferred step rate. The participant will also receive a training log, but will track their pace and distance for each run.

Every participant will perform a 2-3 minute running session on the treadmill after data collection in order to acclimate looking down at the watch, periodically, for 3-5 seconds. This should minimize risk with falling while intermittently looking at the watch for feedback while running overground without supervision.

Volunteers will return after 10 in-field training sessions using their monitoring device and a subset of the study participants will return at 6 months to re-assess AVLR and step rate. The intake questionnaire asks if a participant will remain in the Fort Sam Houston area for 7 months after study enrollment. If the participant mark yes, investigators will ask them if the participant would return for a six month follow-up. Investigators will have 30 runners (15 from control group and 15 from retraining group) return for a six month follow-up.

The watch has GPS capability to provide accurate feedback on the runner's pace and distance. Investigators will not be monitoring GPS location information for the purpose of this study. All running data will be deleted off the watch when the participant return for their follow-up after the 10 in-field training sessions.

A retrospective medical record review, using AHLTA, querying lower extremity injury diagnoses and low back pain will be conducted at six months and at the completion of one year after the retraining program. All volunteers will also receive four email surveys over the year asking them to give their weekly running mileage and (yes/no) if the participant has limited activity due to a running-related overuse injury for one or more days during that quarter. If the answer is yes, the runner will receive additional questions regarding the location and nature of the injury. This quarterly survey is necessary to maximize the accuracy of mileage and injury information to account for mileage conducted and for injuries for which the runner does not seek medical attention. If after 4 weeks the email response rate is less than 50%, the subjects will be contacted by phone to respond to the survey questions. A retrospective profile review, using MODS/Eprofile, querying limited duty days from running-related injuries will be conducted at six months and at the completion of one year after the retraining program. The participants will be required to return the Garmin Watch at the completion of the retraining program or if the participant chooses to leave the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18 - 50 years
* Active Duty, Department of Defense beneficiaries
* History of running-related overuse, musculoskeletal injury of the lower extremity (knee, hip, lower leg, or bone stress injury) within the last six months
* Currently able to run continuously for at least 15 minutes at self-selected pace, 3 times per week.
* Read and speak English well enough to provide informed consent and follow study instructions

Exclusion Criteria:

* Known pregnancy currently or in the previous 6 months
* Lower extremity or low back surgery in the previous 6 months
* Any lower extremity or low back exercise profile that limits running
* Participant has already completed a step rate, gait retraining program
* Participant has a step rate greater than 176 steps per minute

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Average vertical loading rate (AVLR) | Baseline, 10 weeks, 6 months
  The slope of the line on a ground reaction force curve from initial contact to the impact peak
Change in Step rate (SR) | Baseline, 10 weeks, 6 months
  The number of steps a participant takes per minute of running
Injury | 1 year
  The number of lower extremity, over-use injuries sustained within 1 year after completing the ten in-field training sessions

SECONDARY OUTCOMES:
Absolute risk reduction | 1 year
  Change in risk for lower extremity, over-use injuries in those that complete step rate retraining
Limited duty days | 1 year
  Number of days a soldier is non-deployable due to a lower extremity, over-use injury

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heiderscheit BC, Chumanov ES, Michalski MP, Wille CM, Ryan MB. Effects of step rate manipulation on joint mechanics during running. Med Sci Sports Exerc. 2011 Feb;43(2):296-302. doi: 10.1249/MSS.0b013e3181ebedf4. PMID 20581720
- [Background] Willson JD, Ratcliff OM, Meardon SA, Willy RW. Influence of step length and landing pattern on patellofemoral joint kinetics during running. Scand J Med Sci Sports. 2015 Dec;25(6):736-43. doi: 10.1111/sms.12383. Epub 2015 Jan 14. PMID 25585589
- [Background] Lenhart R, Thelen D, Heiderscheit B. Hip muscle loads during running at various step rates. J Orthop Sports Phys Ther. 2014 Oct;44(10):766-74, A1-4. doi: 10.2519/jospt.2014.5575. Epub 2014 Aug 25. PMID 25156044
- [Background] Willy RW, Buchenic L, Rogacki K, Ackerman J, Schmidt A, Willson JD. In-field gait retraining and mobile monitoring to address running biomechanics associated with tibial stress fracture. Scand J Med Sci Sports. 2016 Feb;26(2):197-205. doi: 10.1111/sms.12413. Epub 2015 Feb 4. PMID 25652871